## Addressing Obesity in Early Care and Education Settings

NCT04140032

April 5, 2025

## **Preschool Project Statistical Analysis Plan**

The primary effectiveness outcome was child BMI z-score, calculated from child height and weight measurements using CDC 2000 age- and sex-specific growth charts. We used linear mixed effects models with BMI z-score as the dependent variable; intervention group indicator, time, intervention group-bytime interaction as independent variables; and random effects for school, family (to account for siblings) and child. The intervention effect was tested as a difference in change over time between groups (group-by-time interaction), using alpha of 0.05 two-sided, and scaled to correspond to a 10-month time interval.